CLINICAL TRIAL: NCT06555562
Title: Activating the Cholinergic Anti-Inflammatory Pathway With Focused Ultrasound Stimulation in Healthy Volunteers and People With Inflammatory Arthritis
Brief Title: Activating the Cholinergic Anti-Inflammatory Pathway in Healthy Volunteers and People With Inflammatory Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Surf Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SURF_CLN_002
Record Dates: First submitted 2024-08-03; First posted 2024-08-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Psoriatic Arthritis; Rheumatoid Arthritis; Ankylosing Spondylitis
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis, Rheumatoid; Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Participants will receive active treatment during the visit. There will be a total of 5 visits involving ultrasound, with 2 being a sham and 3 being active. Patient is blinded to the treatment. The visit in which the sham is administered will be determined according to the Randomization Table
  Interventions: Device: Ultrasound Stimulation
- Control (Sham Comparator): Participants will receive a non-active treatment during the visit. There will be a total of 5 visits involving ultrasound, with 2 being a sham and 3 being active. Patient is blinded to the treatment. The visit in which the sham is administered will be determined according to the Randomization Table
  Interventions: Device: Non-active ultrasound stimulation

INTERVENTIONS:
Device: Ultrasound Stimulation — Ultrasound therapy will be administered to the appropriate target.
  Arms: Treatment
Device: Non-active ultrasound stimulation — Non-active ultrasound therapy will be administered to the appropriate target
  Arms: Control

SUMMARY:
This study is designed to investigate whether non-invasive ultrasound (US) that is optimized for stimulation and can elicit an anti-inflammatory response in people with Inflammatory Arthritis as compared to a sham intervention. The primary endpoint is the change in pro-inflammatory cytokines in blood drawn before and after US. Each participant receives 4 experimental US sessions, one of which is randomly assigned to be placebo.

DETAILED DESCRIPTION:
The CAP has demonstrated potential as a treatment for various autoimmune and inflammatory disorders, including inflammatory arthritis (Rheumatoid Arthritis, Psoriatic Arthritis, Ankylosing Spondylitis) and Inflammatory Bowel Disease (Ulcerative Colitis and Crohn's Disease).

The target populations for this study include healthy volunteers and individuals aged 22-75 years diagnosed with Rheumatoid Arthritis (RA), Psoriatic Arthritis (PsA) or Ankylosing Spondylitis (AS) by a board-certified rheumatologist.

Up to 20 healthy volunteers and 40 individuals with RA or PsA will be enrolled. After an initial blood draw, participants will receive either active or sham ultrasound during each visit. There will be a total of 5 visits involving ultrasound, with 2 being a sham and 3 being active. The visit in which the sham is administered will be determined according to the Randomization Table. To ensure participant safety, the ultrasound parameters used for the active sessions will not exceed the FDA's limits.

After the US is completed, participants should be asked to wait in the clinic for a few hours following the completion of the US intervention, after which they will have a second blood draw. Once the second blood draw is completed, participants may leave and resume their regular diet. Participants will be asked to return after 24 hours of their intervention for their third blood draw.

ELIGIBILITY:
Healthy Volunteer Population

Inclusion Criteria:

* 22-75 years of age
* Weigh at least 40 kg

Exclusion Criteria:

* Any physical disabilities, conditions, or diseases that limit the capacity to participate in study procedures or increase the risk of harm as determined by the study PI
* Unable to provide informed consent
* Active bacterial or viral infection
* Class II obesity with a BMI of 35 or higher
* Pregnant women or those trying to become pregnant
* Active use of tobacco/nicotine products
* History of substance use disorder or active regular use of substances (nicotine, marijuana, cocaine, psychedelics, stimulants, etc.)
* Splenomegaly, asplenia, or splenectomy

Inflammatory Arthritis Population

Inclusion Criteria:

* 22-75 years of age
* Weigh at least 40 kg
* Diagnosis of Rheumatoid Arthritis, Psoriatic Arthritis, or Axial Spondyloarthritis of at least 6 months duration as defined by ACR guidelines
* Able to continue the same stable dose of immunomodulatory medication(s) while participating in the study

Exclusion Criteria:

* Unable to provide informed consent
* Took a JAK inhibitor within the last 4 weeks, or likely to start one while participating in this study
* Started a conventional synthetic DMARD (csDMARD) within the last 8 weeks or had a change in prescription within the last 4 week
* Started a Tumor Necrosis Factor (TNF) inhibitor within the last 5 months or had a change in prescription within the last 3 months
* Started any other biologic or targeted synthetic DMARD within the last 3 months, or likely to start one while participating in the study
* Started a corticosteroid, had a change in prescription, or on a stable dose = or > 10 mg of prednisone daily within the last 4 weeks
* Regular use of epinephrine like medications (cold, cough, congestion, or sinus medications, bronchodilators, appetite suppressants)
* Active use of tobacco/nicotine products
* History of substance use disorder or likely use of substances during the study period (marijuana, opioids/heroin, cocaine, psychedelics, methamphetamine, etc.)
* Active bacterial or viral infection
* Receiving chemotherapy or immunotherapy to treat malignancy
* Significant immunodeficiency due to underlying illness
* Class II obesity with a BMI of 35 or higher
* Pregnant women or those trying to become pregnant
* Wound, rash, infection, or traumatic injury over the target area
* Vagal nerve injury or vagotomy
* Surgery or major traumatic injury in the past 90 days
* Chronically-implanted medical devices (i.e. pacemaker, AICD, vagus nerve stimulator, spinal cord stimulator)
* Clinically significant cardiovascular disease
* CKD Stage 3 or higher
* Uncontrolled fibromyalgia or other diffuse pain syndromes

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Tumor Necrosis Factor Alpha Concentration Differences | Baseline to 2 hours post therapy
  Measure the change before and after ultrasound stimulation by immunoassay of blood plasma after challenge with LPS.

SECONDARY OUTCOMES:
Interleuken 1b Concentration Difference | Baseline to 2 hours and 24 hours post therapy
  Measure the change before and after ultrasound stimulation by immunoassay of blood plasma after challenge with LPS.
Interleuken IL-6 Concentration Difference | Baseline to 2 hours and 24 hours post therapy
  Measure the change before and after ultrasound stimulation by immunoassay of blood plasma after challenge with LPS.
Tumor Necrosis Factor Alpha Concentration Differences | Baseline to 24 hours post therapy
  Measure the change before and after ultrasound stimulation by immunoassay of blood plasma after challenge with LPS.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tekton Research, Austin, Texas
  - UT Health, Houston, Texas

IPD SHARING:
Plan to Share IPD: No